CLINICAL TRIAL: NCT01791959
Title: The Effects of Synbiotics Supplement on Lipid Profile, Liver Enzymes, Inflammatory Factors and Hepatic Fibrosis in Patients With Nonalcoholic Steatohepatitis
Brief Title: The Effects of Synbiotics Supplement on Biochemical Factors and Hepatic Fibrosis in Patients With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 046466
Record Dates: First submitted 2013-02-05; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Synbiotic (Active Comparator): 2 synbiotic capsules for 28 weeks
  Interventions: Dietary Supplement: synbiotic
- maltodexterin (Placebo Comparator): two capsules per day for 28 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: synbiotic — 2 symbiotics capsules per day for 28 weeks
  Arms: Synbiotic
Other: placebo — 2 Maltodexterin capsules as a placebo per day for 28 weeks
  Arms: maltodexterin

SUMMARY:
To study the effects of synbiotics supplement on lipid profile, liver enzymes, inflammatory factors and hepatic fibrosis in patients with Nonalcoholic Steatohepatitis (NASH), 50 patients who referred to Gastrointestinal (GI) clinic with steatosis grade 1 or more will be randomly allocated to receive 2 protexin capsules or placebos for 7 months; both groups will be advised to adherence our diet and exercise program too. At the first and the end of the intervention, lipid profiles, liver enzymes, some inflammatory cytokines, and liver fibrosis will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 70 years
* Body Mass Index (BMI) between 25-40
* Serum alaninaminotransferase more than 1.5 fold of upper limit of normal range
* Sonographic findings compatible with hepatic steatosis (degree 2 or more)

Exclusion Criteria:

* Diabetes
* Taking any kind of antibiotics two weeks before recruitment
* History of alcohol consumption
* pregnancy or lactation
* Professional athletes
* Other liver disease (viral/etc)
* Use of drugs such as calcium channel blockers, high dose synthetic estrogens, methotrexate , amiodarone, steroids, chloroquine, immunosuppressive drugs, lipid-lowering agents, metformin and vitamin E
* A history of Hypertension, Cardiovascular disease, Pulmonary disease, Renal disease & Celiac disease; Cirrhosis
* History of Upper GI surgery / Prior surgical procedures such as jejunoileal or jejunocolic bypass, gastroplasty
* Following program to lose weight in recent 3 mo
* A history of hypothyroidism or Cushing's syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Alaninaminotransferase (ALT) | 28 weeks
Liver fibrosis | 28 weeks

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Azita Hekmatdoost, MD, PhD, Principal Investigator — National Nutrition and Food Technology Research Institute

REFERENCES:
- [Derived] Eslamparast T, Poustchi H, Zamani F, Sharafkhah M, Malekzadeh R, Hekmatdoost A. Synbiotic supplementation in nonalcoholic fatty liver disease: a randomized, double-blind, placebo-controlled pilot study. Am J Clin Nutr. 2014 Mar;99(3):535-42. doi: 10.3945/ajcn.113.068890. Epub 2014 Jan 8. PMID 24401715